CLINICAL TRIAL: NCT02704351
Title: Retrospective Chart Review of Fast-track Cardiac Anesthesia Using Suggamadex for Rapid Reversal of Neuromuscular Blockade Following Cardiac Surgery in a Developing Country
Brief Title: Suggamadex and Fast-track Cardiac Anesthesia in a Developing Country
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-01162
Record Dates: First submitted 2016-03-04; First posted 2016-03-10 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Suggamadex; Surgery for Congenital Heart Disease
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sugammadex group: sugammadex to reverse neuromuscular blockade following cardiac surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Sugammadex to reverse neuromuscular blockade

SUMMARY:
The purpose of this study is to retrospectively review our preliminary experience during a surgical trip to Tuxtla, Mexico, using suggamadex to reverse neuromuscular blockade following CPB and cardiac surgery for repair of CHD in infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent cardiac surgery and cardiopulmonary bypass in Tuxtla, Mexico in September 2015.

Exclusion Criteria:

* None

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Last September 2015, patients in Tuxtla, Mexico who underwent cardiac surgery and cardiopulmonary bypass surgery for congenital heart defect where suggamadex was used for reversal of neuromuscular blockade.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Clinical effects of the reversal of neuromuscular blockade with suggamadex following surgery for congenital heart disease in infants and children | After cardiac surgery, on average within 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided